CLINICAL TRIAL: NCT02734485
Title: The Use of Deep TMS for the Treatment and Rehabilitation of Patients With Parkinson's Disease and Progressive Supranuclear Palsy
Brief Title: Deep TMS for the Treatment of Patients With Parkinson's Disease and Progressive Supranuclear Palsy
Acronym: DeepTMSPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RP 16/13
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Progressive Supranuclear Palsy; Parkinson's Disease
Keywords: Progressive supranuclear palsy; Deep transcranial magnetic stimulation
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active Deep Tms (Active Comparator): Each DTMS session consisted in two consecutive stimulations: a first low-frequency (1 Hz) stimulation in the motor cortex (110% of the motor threshold, for 15 minutes)and a second high-frequency (10Hz) one in the prefrontal cortex (100% motor threshold, 2 seconds each train, 20 seconds between trains, for 15 minutes).The coil contains two symmetric devices, perfectly designed to rouse both hemispheres at the same time.
  Interventions: Device: active Deep TMS
- sham deep tms (Sham Comparator): The Sham DTMS consisted in the same protocol of active treatment with the same preparation of the subject and settings of the instrument but with an inactive DTMS coil.
  Interventions: Device: sham Deep TMS

INTERVENTIONS:
Device: active Deep TMS — The Brainsway DTMS produces a time-varying magnetic field and, based on Faraday's Law, it can be assumed that a time-varying magnetic field generates an electrical current in a nearby conductive substance. The induced electric current in the cortex travels in an orthogonal path in the direction of the magnetic field with the maximum strength and current located beneath the coil in the helmet placed on the patient's head and transmits magnetic pulses to the patient's brain. The induced current is tangential to the scalp at the cortical surface, and decreases in magnitude with increasing depth.
  Patients underwent 12 sessions, 3 times a week, of repetitive DTMS using the novel H2-coil (Brainsway LDT).
  Arms: active Deep Tms
Device: sham Deep TMS — The Sham DTMS consisted in the same protocol of active treatment with the same preparation of the subject and settings of the instrument but with an INACTIVE DTMS coil.
  Arms: sham deep tms

SUMMARY:
Background: Progressive supranuclear palsy (PSP) is a rare neuro-degenerative disease, counted among atypical parkinsonism (AP). Medical treatment and rehabilitation are extremely limited in AP, therefore it would be very useful to find new ways to improve motor and non motor symptoms in PSP. The Brainway Deep Transcranial magnetic stimulation (DTMS) is a new technology of TMS using a particular coil, i.e. H-coil, able to stimulate deeper regions of the brain. Only few studies in literature have evaluated the efficacy of DTMS in Parkinson's Disease and parkinsonism; in particular in PSP patients, a case report showed an improvement in language.

DETAILED DESCRIPTION:
Materials and Methods: This study was a pilot, randomized, cross-over, double blind trial. It was designed to evaluate the efficacy of Deep TMS in terms of recovery of motor functions, freezing of gait, and cognitive decline in patients with PSP. Nineteen subject underwent 14 session of high frequency DTMS over a 4 weeks period. The target were the left Broca and dorsolateral prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with PSP according to NINDS-SPSP criteria

Exclusion Criteria:

* contraindications for DTMS (history of seizures, pacemakers, or any other electric device)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in PSP rating scale total score between baseline evaluations (T0 orT2) and end of treatment (T1 or T3) | evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation (after four weeks of treatment): T1 for first period, T3 for second period).
  Clinical measures were summarized as means and standard deviations for all the 19 patients and stratified by treatment (active and sham) and evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation: T1 for first period, T3 for second period).

SECONDARY OUTCOMES:
Change in MoCA total score between baseline evaluations (T0 orT2) and end of treatment (T1 or T3) | evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation (after four weeks of treatment): T1 for first period, T3 for second period
  Clinical measures were summarized as means and standard deviations for all the 19 patients and stratified by treatment (active and sham) and evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation: T1 for first period, T3 for second period).
Change in PDQ 39 total score between baseline evaluations (T0 orT2) and end of treatment (T1 or T3) | evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation (after four weeks of treatment): T1 for first period, T3 for second period
  Clinical measures were summarized as means and standard deviations for all the 19 patients and stratified by treatment (active and sham) and evaluation time
Change in NMS total score between baseline evaluations (T0 orT2) and end of treatment (T1 or T3) | evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation (after four weeks of treatment): T1 for first period, T3 for second period
  Clinical measures were summarized as means and standard deviations for all the 19 patients and stratified by treatment (active and sham) and evaluation time
Change in Hamilton rating scale for depression total score between baseline evaluations (T0 orT2) and end of treatment (T1 or T3) | evaluation time (pre-stimulation: T0 for first period, T2 for second period; post-stimulation (after four weeks of treatment): T1 for first period, T3 for second period
  Clinical measures were summarized as means and standard deviations for all the 19 patients and stratified by treatment (active and sham) and evaluation time

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Stocchi, MD, PHD, Principal Investigator — IRCCS SAN RAFFAELE PISANA
Locations (1):
- Irccs San Raffaele Pisana, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Boeve BF. Progressive supranuclear palsy. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1:S192-4. doi: 10.1016/S1353-8020(11)70060-8. PMID 22166432
- [Background] Levkovitz Y, Roth Y, Harel EV, Braw Y, Sheer A, Zangen A. A randomized controlled feasibility and safety study of deep transcranial magnetic stimulation. Clin Neurophysiol. 2007 Dec;118(12):2730-44. doi: 10.1016/j.clinph.2007.09.061. Epub 2007 Oct 30. PMID 17977787
- [Background] Trebbastoni A, Raccah R, de Lena C, Zangen A, Inghilleri M. Repetitive deep transcranial magnetic stimulation improves verbal fluency and written language in a patient with primary progressive aphasia-logopenic variant (LPPA). Brain Stimul. 2013 Jul;6(4):545-53. doi: 10.1016/j.brs.2012.09.014. Epub 2012 Oct 24. PMID 23122915
- [Derived] Radicati FG, Vacca L, Casali M, Tremigliozzi I, Alborghetti M, Lombardi M, Rossini PM, Stocchi F. Deep transcranial magnetic stimulation in progressive supranuclear palsy: a randomized double-blind, cross-over study. Neurol Sci. 2025 Dec;46(12):6923-6931. doi: 10.1007/s10072-025-08549-1. Epub 2025 Nov 12. PMID 41219570